CLINICAL TRIAL: NCT03304808
Title: A Randomized, Controlled Study of the Efficacy of a New Behavioral Treatment for Premature Ejaculation Using a Masturbation Aid Device
Brief Title: Efficacy of a New Behavioral Treatment for Premature Ejaculation Using a Masturbation Aid Device: Star-Stop 3.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Sexológico Murciano (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISMSEXOLOGIA
Record Dates: First submitted 2017-03-30; First posted 2017-10-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Premature Ejaculation; Cognitive-Behavior Treatment; Masturbation Aid Device
Keywords: premature ejaculation; cognitive-behavior; treatment; device
MeSH Terms: conditions — Premature Ejaculation | interventions — Lubricants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- device (Experimental)
  Interventions: Device: Exercise Programme +device+ lubricant
- behavioral (Active Comparator)
  Interventions: Behavioral: Exercise Programme + lubricant
- waiting list (No Intervention)

INTERVENTIONS:
Device: Exercise Programme +device+ lubricant — A first line treatment for the PE of a new 7 weeks exercise programme to control male orgasm using a masturbation aid device in a variation of the classical stop-start technique first introduced by Semans in 1956.
  Four exercise:
  1. Exercise of Masturbation that intends to raise awareness of the ejaculatory response and identify the tension on the muscles of the genital area .
  2. Star and Stop to identify the tension and try to reduce this tension, on the pelvic floor muscles pay special attention to the anal sphincter.
  3. Delay the ejaculatory response on four different occasions, by loosening the tension in the genital area and relaxing the anal sphincter not stop masturbating
  4. Practice the ability to delay ejaculation as in previous exercises, but this time performing hip movements similar to penetration not stop masturbating
  Arms: device
Behavioral: Exercise Programme + lubricant — A first line treatment for the PE of a new 7 weeks exercise programme to control male orgasm using a masturbation aid device in a variation of the classical stop-start technique first introduced by Semans in 1956.
  Four exercise:
  1. Exercise of Masturbation that intends to raise awareness of the ejaculatory response and identify the tension on the muscles of the genital area .
  2. Star and Stop to identify the tension and try to reduce this tension, on the pelvic floor muscles pay special attention to the anal sphincter.
  3. Delay the ejaculatory response on four different occasions, by loosening the tension in the genital area and relaxing the anal sphincter not stop masturbating
  4. Practice the ability to delay ejaculation as in previous exercises, but this time performing hip movements similar to penetration not stop masturbating
  Arms: behavioral

SUMMARY:
The present study included 57 patients ≥18 years who met diagnostic criteria for PE including intravaginal ejaculatory latency time (IELT) of ≤2 minutes and had a Premature Ejaculation Diagnostic Tool (PEDT) score ≥11.

Subjects were randomized to an experimental group that used the device with exercise programme (n=18) a first control group that only used the exercise programme (n=17) and a wait-list control group (n=22).

As a main outcome measure used stopwatch-measured average IELT, Premature Ejaculation Profile (PEP), and the Golombok-Rust Inventory of Sexual Satisfaction (GRISS).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be heterosexual males
* To be in a stable monogamous, sexual relationship with a female partner for at least 6 months,
* Must score = 11 in the Premature Ejaculation Diagnostic Tool (PEDT).
* Must have a self-estimated average intravaginal ejaculatory latency time (IELT) of <2 min. -Must be in good general health with no clinically significant abnormalities as determined by medical history and clinical lab results.

Exclusion Criteria:

* To suffer an alteration or mental disorder according to the criteria of the DSM-IV.
* History of alcohol abuse and dependence.
* Do not to consume medication, drugs of recreative use or alcohol (except for caffeine or nicotine/tobacco).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
IELT FOLD INCREASE | 7 weeks
  fold changes are defined directly in terms of ratios.If the initial value is A and the final value B, the fold change is defined as B/A

SECONDARY OUTCOMES:
Premature Ejaculation Profile (PEP) | 7 weeks
  proportion of patients who achieved criteria for clinical benefit, defined as achieving a two-category or greater increase in the change in control over ejaculation and level of satisfaction with intercourse, and a one-category or greater increase in the change in ejaculation-related distress and degree of interpersonal difficulty.

OTHER OUTCOMES:
Golombok Rust Inventory of Sexual Satisfaction (GRISS) | 7 weeks
  Scale ejaculatory function

CONTACTS AND LOCATIONS:
Locations (1):
- Jesús Rodríguez, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided